CLINICAL TRIAL: NCT05248035
Title: Automated Pupillometry and Delirium in Patients on Mechanical Ventilation in Intensive Care-intensive Care
Brief Title: PupillOmetry for Prediction of DelirIUM
Acronym: PODIUM
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201165; 2020-A03517-32 (Other: IDRCB)
Record Dates: First submitted 2021-12-09; First posted 2022-02-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Delirium; ICU
Keywords: Automated Pupillometry Delirium ICU
MeSH Terms: conditions — Delirium | interventions — Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Adult patient hospitalized in ICU for a duration of mechanical ventilation longer than 48 hours
  Interventions: Other: Adult patient hospitalized in ICU

INTERVENTIONS:
Other: Adult patient hospitalized in ICU — acquisition of dynamic parameters in addition to pupillary diameter, such as . pupillary diameter, variation of the pupillary diameter, pupillary constriction speed, pupillary dilatation speed, photomotor reflex latency, NPi and symmetry of pupillary responses after a standardized light stimulus

SUMMARY:
Delirium in intensive care unit (ICU) is a serious event. It is associated with short-term complications (agitation, self-extubation, accidental removal of catheters, prolonged length of stay and ventilation), excess mortality, functional and cognitive impairment. It is particularly frequent in patients requiring mechanical ventilation but diagnosis is not easy. There are screening scales, but it is insufficiently used in clinical practice: Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) or Intensive Care Delirium Screening Checklist (ICDSC). These scales are time consuming and require trained personnel. Automated pupillometry (AP) is a new device to objectively, rapidly, and reproducibly identify acute brain dysfunction. Recent data suggest that AP could be used to predict delirium in the ICU. This would need to be validated for routine use in the ICU.

Evaluate AP parameters on day 3 of invasive mechanical ventilation as a predictive tool for CAM-ICU diagnosed delirium during the first 14 days of ICU stay.

Study design: Prospective, multicenter, non-interventional cohort

Measurement of the AP parameters at day 3 after ICU admission and their predictive performance for delirium: pupillary diameter, variation of the pupillary diameter, pupillary constriction speed, pupillary dilatation speed, photomotor reflex latency, NPi and symmetry of pupillary responses.

DETAILED DESCRIPTION:
Automated pupillometry is an easy-to-use device that allows for accurate objective assessment of the photomotor reflex.

AP it allows the acquisition of dynamic parameters in addition to pupillary diameter, such as quantitative measurement of pupillary reactivity, speed, or latency of pupil contraction after a standardized light stimulus.

Automated pupillometry has been evaluated in ICU, in a monocentric study in non-brain-damaged patients, AP was used for the first time to predict the occurrence of delirium. Interestingly, the decrease in pupillary diameter variation at day 0 after 48h of IMV (D0) was independently associated with the occurrence of delirium during the ICU stay. This seems promising but requires a validation study in order to recommend its routine use.

The hypothesis is the AP parameters predict the risk of delirium in ICU-patients ventilated for more than 48 hours. Specifically, AP parameters on the D3 of mechanical ventilation allow predicting the occurrence of delirium during the first 14 days of resuscitation. This will allow early change of patient management, by identifying patients at risk of delirium and serious short-term adverse events.

This is a prospective, observational, multicenter cohort study involving 5 ICU in the Paris area.

To ensure the 213 planned inclusions and the 3-month follow-up of all included patients, a research duration of 15 months is expected. The ethical committee of the French Society of intensive care medicine (FICS) approved the study protocol (CE SRLF 20-09) and required Family members' informed consent.

At D0, patient is included and we start to evaluate AP parameter twice a day from D0 to D7 and to monitor delirium occurrence using Confusion assessment monitoring in the ICU (CAM ICU).

We assess changes in AP parameters from D0 to D7 of mechanical ventilation in patients with and without CAM-ICU diagnosed delirium during the first 14 days of ICU stay.

Automated pupillometry protocol : The AP is measured for each eye from D0 onwards, twice a day, as long as the patient is under mechanical ventilation and up to a maximum of 7 days (D7), using the NPI Neuroptics® device. These parameters were measured by the nurses or by the investigating physician not involved in the patient's care. At each measurement point, the mean value of both eyes was used for the analyses. The AP parameters are: pupillary diameter, variation of the pupillary diameter, pupillary constriction speed, pupillary dilatation speed, photomotor reflex latency, NPi and symmetry of pupillary responses. Routine neurological monitoring in ICU includes the RASS score every 4 hours. If the RASS score is ≥ -3 then CAM-ICU will be administered twice daily starting on day 3 by the patient's attending physicians. The physicians in charge of the patient will be blinded to the AP results.

ELIGIBILITY:
Inclusion criteria :

* Adults ≥ 18 years
* mechanical ventilation since 48h
* Information and no opposition of patient or close person if he is present at the time of inclusion, otherwise urgent inclusion

Exclusion criteria :

* Patient diagnosed confused by CAM-ICU on D0
* Ophthalmological pathology modifying the photomotor reflex
* Acute or chronic neurological pathology: Cerebro-injured patients (head trauma, stroke, cardiopulmonary arrest, hypoglycemic coma, meningitis / encephalitis / brain abscess), dementia with MMSE <24
* Duration of stay in intensive care> 72h or duration of ventilation> 72h
* Readmission in intensive care
* Moribund patient
* Patient under guardianship or curatorship
* No affiliation to social security (beneficiary or assignee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient hospitalized in ICU for a duration of mechanical ventilation longer than 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Measurement of the parameters of the automated pupillometry | at day 0

SECONDARY OUTCOMES:
Measurement of the parameters of the automated pupillometry | until 7 days
Rate of agitated patients (agitation is defined by a Richmond Agitation-Sedation Scale > +1(RASS score: +4; -5 with 0= better outcome) requiring use of neuroleptics or dexmedetomidine) | until day14 of resuscitation or discharge from resuscitation
Self-extubation rate | until day14 or stop invasive ventilation
Accidental catheter ablation rate | up to day14 resuscitation or resuscitation discharge
Number of days of mechanical ventilation | until D14 or stopping invasive ventilation
Number of days in intensive care | until day90
Death rate | at day90
Early PREdiction of DELIRium in ICu patients (E-PRE-DELIRIC) score | at day 0
Measurement of the parameters of the automated pupillometry in the subgroup of patients hospitalized for sepsis | day0
Measurement of the parameters of the automated pupillometry in the subgroup of patients hospitalized for cardiogenic shock under veno-arterial circulatory support | day0

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Jaquet, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat-Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jaquet P, Couffignal C, Tardivon C, Godard V, Bellot R, Assouline B, Benghanem S, Da Silva D, Decavele M, Dessajan J, Hermann B, Rambaud T, Voiriot G, Sonneville R; PODIUM Study Group. PupillOmetry for preDIction of DeliriUM in ICU (PODIUM): protocol for a prospective multicentre cohort study. BMJ Open. 2023 Jul 12;13(7):e072095. doi: 10.1136/bmjopen-2023-072095. PMID 37438060